CLINICAL TRIAL: NCT05793398
Title: Pathomechanisms in Patients With Cardiac Sarcoidosis and Other Inflammatory and Familial Cardiomyopathies of Similar Phenotypic Appearance
Brief Title: Biomaterial Collection - and Analysis in Cardiac Sarcoidosis
Status: Not yet recruiting | Type: Observational
Sponsor: Heart Center Leipzig - University Hospital (Other)
Collaborators: University of Leipzig Medical Center, Department of Cardiology (Unknown); Heart and Diabetes Center North Rhine-Westphalia, Erich and Hanna Klessmann Institute for Cardiovascular Research and Development (Unknown); Max Delbrück Center for Molecular Medicine (MDC), Berlin (Unknown)
Responsible Party: Sponsor
Other Study IDs: CD1022
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endomyocardial biopsy-positive Cardiac sarcoidosis
- Endomyocardial biopsy-negative non ischemic cardiomyopathy

SUMMARY:
Cardiac sarcoidosis (CS) is a complex disease that is characterized by the formation of inflammatory granulomas in the myocardium. The exact underlying pathophysiology of the disease is not yet fully understood, but it is believed to be related to dysregulation of the immune system. Despite significant progress in recent years, the disease remains difficult to diagnose, and there is a high risk of severe complications such as life-threatening cardiac arrhythmias, severe heart failure, and sudden cardiac death in affected patients.

Moreover, the clinical presentation of CS can be similar to other inflammatory heart diseases or familial cardiomyopathies. Thus, it is challenging to differentiate between these diseases, which can lead to a delayed diagnosis and poor prognosis. It is unclear whether certain genetic variants play a role in the clinical course and prognosis of CS, which highlights the need for more research in this area.

The diagnosis of CS requires cardiac or extracardiac biopsy with granuloma detection, which is an invasive and complex procedure. Consequently, the disease is thought to be underdiagnosed, and many affected patients may not receive timely treatment, resulting in excess mortality. Early diagnosis and immunosuppressive treatment, as well as defibrillator implantation if necessary, are crucial in delaying disease progression, preventing complications, and improving prognosis.

To better understand the key molecular pathological mechanisms underlying the development and maintenance of CS, a prospective, multicenter, exploratory study has been initiated. The project involves the collection, storage, and analysis of biological samples from blood, myocardium, and lymph nodes of patients with cardiac sarcoidosis or cardiomyopathies that present clinically and image morphologically similar. The samples will be used for scientific investigations on disease mechanisms of cardiomyopathies as well as for identification of new biomarkers in cardiomyopathy diagnostics and for follow-up of therapeutic measures.

The study will employ a range of classical biochemical methods such as ELISA, RIA, as well as more modern methods of molecular biology (single cell sequencing, single nucleus sequencing) and systems biology (genomics, metabolomics, or proteomics) to identify key molecular pathological mechanisms in the development and maintenance of CS.

In addition, genetic analysis will be performed to investigate cardiomyopathy- and ion channel-associated genetic variants, which is critical for improving diagnostics and early, individualized therapy. The study will be conducted on a multicenter basis, with the Heart Center Leipzig serving as the initiator and lead center and the University Hospital Leipzig as the second study center. Biochemical and molecular biological analyses will be performed on behalf of the study management at the Heart Center Leipzig, the University Hospital Leipzig, and the Erich and Hanna Klessmann Institute for Cardiovascular Research and Development of the Heart and Diabetes Center NRW and Max Delbrück Center for Molecular Medicine in Berlin.

In conclusion, CS is a complex and challenging disease that requires further research to better understand its underlying mechanisms and improve diagnostic and therapeutic strategies. The prospective, multicenter, exploratory study will provide valuable insights into the disease's key molecular pathological mechanisms and identify new biomarkers for better diagnostics and individualized therapy.

ELIGIBILITY:
Inclusion Criteria:

(a) patients with a history of symptomatic cardiac sarcoidosis/inflammatory cardiomyopathy or b) patients with newly diagnosed heart failure with cardiac arrhythmias (ventricular tachycardia, conduction disturbances, etc.) that may indicate sarcoidosis or inflammatory cardiomyopathy or c) patients with image morphological suspicion of cardiac sarcoidosis or inflammatory cardiomyopathy (MRI, PET-CT) or (d) patients who require or have received a ventricular assist device (VAD) or cardiac transplantation due to suspected cardiac sarcoidosis or inflammatory cardiomyopathy and (e) written informed consent has been obtained from patients for study participation and consent for analysis of patient samples. Studies on pseudoanonymized samples will only be performed with appropriately signed informed consent.

Exclusion Criteria:

1. Patients with psychiatric illness that impairs business or insight capacity.
2. Patients with chronic heart failure due to coronary artery disease or valvular vitiation.
3. severe underlying disease other than sarcoidosis that is likely to result in death within one year.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic patients with suspected inflammatory cardiomyopathy and/or conduction disorders and/or ventricular arrhythmias, suspected cardiac sarcoidosis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
CD14++CD16+ - monocytes/macrophages in myocardial samples and peripheral blood correlates with disease activity | Baseline
  Sarcoidosis leads to a cellular TH1-mediated immune response with formation of non-necrotizing granulomas in affected organs, including the heart. Monocyte/macrophage subpopulations play an important role in the initiation of the TH1 immune response. Detection of specific immune cells such as CD14++CD16+ - monocytes/macrophages in myocardial samples and peripheral blood correlates with disease activity.
Specific genetic variants, single nucleotide polymorphisms, and epigenetic markers are associated with an individually increased risk of disease. | Baseline
  Modern genetic testing methods can detect an individually increased risk of disease.

IPD SHARING:
Plan to Share IPD: No